CLINICAL TRIAL: NCT01778283
Title: Comparison of Cardiac Index and Cardiac Output Effect During Maintenance Hemodialysis Between Acetate-Free and Acetate-Based Online Hemodiafiltration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Khajohn Tiranathanagul, Doctor, Chulalongkorn University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 297/55
Record Dates: First submitted 2012-12-20; First posted 2013-01-29 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: End-stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acetate-free solution first (Experimental): Acetate-free solution first : hemodialysis 4 hours with Acetate-free solution (Acetate 0 mEq/L Citrate 2 mEq/L) at the first session after enrollment, and then switch to Acetate-based solution (Acetate 3 mEq/L Citrate 0 mEq/L) at the next 4-hr hemodialysis session
  Interventions: Biological: Acetate-free dialysis solution
- Acetate-based solution first (Active Comparator): Acetate-based solution first : hemodialysis 4 hours with Acetate-based solution (Acetate 3 mEq/L Citrate 0 mEq/L) at the first session after enrollment, and then switch to Acetate-free solution (Acetate 2 mEq/L Citrate 2 mEq/L) at the next 4-hr hemodialysis session
  Interventions: Biological: Acetate-free dialysis solution

INTERVENTIONS:
Biological: Acetate-free dialysis solution — the hemodialysis solution that does not contain acetate as buffer

SUMMARY:
The purpose of this study is to detemine whether effect of Acetate-free solution on cardiac index and cardiac output measured by saline dilution techniques compares with Acetate-based solution in online-hemodiafiltration

ELIGIBILITY:
Inclusion Criteria:

* End-stage renal disease patients with age over 20 years and stable clinical status
* Dialytic age > 6 months
* Maintenance hemodialysis with online-hemodiafiltration mode at King Chulalongkorn Memorial Hospital
* Use arteriovenous fistula or arteriovenous graft as vascular access for hemodialysis
* No vascular access recirculation
* No liver impairment
* No severe, intractable metabolic acidosis or alkalosis (HCO3 <15, >30)
* No pre-existing severe, intractable hypocalcemia (Ca < 7.5) or clinical of hypocalcemia

Exclusion Criteria:

* On hemodialysis via tunnel catheter
* Vascular access recirculation
* Liver dysfunction
* Severe, intractable metabolic acidosis or alkalosis (HCO3 <15, >30)
* Pre-existing severe, intractable hypocalcemia (Ca < 7.5) or clinical of hypocalcemia
* Acute or recent myocardial ischemia or congestive heart failure (within 1 months)
* Threatening arrhythmia (VT, VF, sustained SVT, AF with rapid ventricular response)
* Patients affected by acute or chronic infections, malignant tumor

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
cardiac index | 6 months
  cardiac index and cardiac output was measured by ultrasound dilution technique
Cardiac output | 6 months
  cardiac index and cardiac output was measured by ultrasound dilution technique

SECONDARY OUTCOMES:
blood pressure | 6 months
peripheral vascular resistance | 6 moths
Patients' symptoms | 6 months
  dizziness, palpitation, nausea, cramp, numbness

OTHER OUTCOMES:
cardiac marker, serum electrolyte, inflammatory marker | January 2013
  BUN, creatinine, serum sodium, serum potassium, serum bicarbonate, serum calcium, ionized calcium, serum magnesium, serum osmol, troponin T, NT-proBNP, CKMB, hs-CRP

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Chulalongkorn University, Bangkok, Bangkok, Thailand